CLINICAL TRIAL: NCT00273754
Title: A Pilot Study to Evaluate if Caffeine Helps Children With Obstructive Sleep Apnea Recover Faster From Anesthesia, and With Less Complications After General Anesthesia for Tonsillectomy and Adenoidectomy.
Brief Title: The Effect of Caffeine on Postextubation Adverse Respiratory Events in Children With Obstructive Sleep Apnea (OSA).
Acronym: OSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC-MS-03-108
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Apnea, Obstructive; Tonsillectomy; Adenoidectomy; Postoperative Complications
Keywords: Obstructive Sleep Apnea (OSA); Tonsillectomy and Adenoidectomy (T&A); Postoperative Complications; Recovery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Postoperative Complications | interventions — Caffeine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo
- Caffeine (Active Comparator): Caffeine benzoate
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Children in group one will receive caffeine benzoate 20 mg/kg i.v., which is equal to a 10 mg/kg caffeine base.
  Arms: Caffeine
Drug: Placebo — Children in group two will receive an amount of normal saline equal to Caffeine
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a research study using caffeine in children who have an obstructive sleep apnea (OSA). OSA means children who stop breathing during their sleep due to obstruction in their airway. The purpose of this study is to determine whether caffeine when given in the vein, will wake children up faster and decrease post-anesthesia airway obstruction, as well as the safety and if the drug agrees with the child compared to a placebo (an inactive or dummy agent).

DETAILED DESCRIPTION:
Patients with OSA are reported to have a higher rate of severe respiratory complications associated with upper airway obstruction during anesthesia and sedation or immediately after anesthesia. Children with OSA (especially those under three years of age, those with severe OSA, cerebral palsy or craniofacial anomalies) are at increased risks for post-operative complications, and require careful monitoring post-operatively.

Although the etiology of obstructive sleep apnea is mainly obstruction due to anatomical and neuromuscular abnormalities, we believe that a central element may contribute to OSA.

The aim of this study is to evaluate whether administration of caffeine to children with OSA, scheduled for elective T & A under general anesthesia contributes to a faster recovery, less post-operative complications, and a shorter stay in the PACU, DSU and the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2.5-18 years old
* Diagnosed with obstructive sleep apnea
* Undergoing elective tonsillectomy and adenoidectomy

Exclusion Criteria:

* Age below 2.5 or above 18 years

Ages: 30 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2003-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samia N. Khalil, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas, Health Science Center at Houston, Children's Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Normal Saline
Period: Overall Study
Arm/Group | Placebo | Caffeine
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Caffeine | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 36 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.3 (2.9) | 5.3 (2.2) | 5.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Who Developed Postextubation Adverse Respiratory Events Compared to Placebo.
Description: The number of children having adverse post-extubation respiratory events, including laryngospasm, upper airway obstruction, apnea, desaturation (defined as decrease in oxygen saturation <95% while breathing oxygen via mask for any length of time) and need for reintubation, both in the Operating Room and in the PACU was recorded.
Time Frame: Time post extubation in OR and PACU until the patient was discharged from the PACU to go home or to a hospital room.
Population: The analysis was per protocol.
Measure: Number; unit: Participants
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 36 | 36
Participants | 21 | 11

2. Secondary Outcome: Occurence of Post Extubatory Respiratory Adverse Events.
Description: The overall occurance of adverse post-extubation respiratory events, including laryngospasm, upper airway obstruction, apnea, desaturation (defined as decrease in oxygen saturation <95% while breathing oxygen via mask for any length of time) and need for reintubation, both in the OR and in the PACU was noted.
Time Frame: Time post extubation in OR and PACU until the patient was discharged from the PACU to go home or to a hospital room.
Population: Per protocol
Measure: Number; unit: Participants
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 36 | 36
Participants | 34 | 17

3. Secondary Outcome: Extubation Time.
Description: Time from end of anesthesia until extubation.
Time Frame: Duration from anesthesia end until extubation time.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 36 | 36
minutes | 11.3 (9.4) | 8.6 (4.9)

4. Secondary Outcome: Awakening Time
Description: A child with a Steward Recovery Scale score of 6 is defined as awake, coughing/crying, and has purposeful movements.
Time Frame: Awakening time from end of anesthesia until the child reached a score of 6 on the Steward recovery score.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 36 | 36
Minutes | 26.6 (16.0) | 26.1 (28.8)

5. Secondary Outcome: Post Anesthesia Care Unit (PACU) Duration
Time Frame: Time spent in PACU following surgical procedure prior to discharge home or hospital admission.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 36 | 36
minutes | 74.4 (43.7) | 84.8 (44.1)

6. Secondary Outcome: Hospital Discharge Time
Description: Children were discharged from the hospital when they reached the hospital discharge criteria: they were awake, had stable vital signs, were breathing adequately, had O2 saturation >95% while breathing room air, were able to swallow fluids, had no or minimal pain, and were able to ambulate without excessive nausea, vomiting, or dizziness.
Time Frame: Total time from end anesthesia to discharge home
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 36 | 36
Minutes | 107.0 (54.5) | 98.2 (55.9)

ADVERSE EVENTS:
Arm/Group | Placebo | Caffeine
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes